CLINICAL TRIAL: NCT05981664
Title: Level Up! Adaptive Gaming for Children With Upper Limb Differences
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Rehabilitation Centre for Children, Canada (Other)
Responsible Party: Principal Investigator, Meghan Guglich, Principal Investigator, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HS25775 (B2022:110)
Record Dates: First submitted 2023-05-09; First posted 2023-08-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Upper Limb Amputation at the Wrist; Pediatric; Upper Limb Amputation; Upper Limb Amputation at the Hand; Amniotic Band Syndrome; Upper Limb Amputation Below Elbow (Injury)
Keywords: pediatric; upper limb difference; one handed gaming
MeSH Terms: conditions — Amniotic Band Syndrome; Wounds and Injuries

STUDY DESIGN:
Masking Description: All participants are provided the intervention, and act as their own control when they are evaluated with and without the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- with adapter (Experimental): All participants are in the experimental group baseline speed and accuracy using minecraft videogame will serve as baseline data and each subject will be their own control. participants will be given an adapter to support onehanded game play and an xbox system to use at home for a week. Follow-up data (speed and accuracy of minecraft) will be reevaluated one week later. Qualitative interview data will assist in understanding facilitators and barriers for use. On baseline and reassessment, the QUEST 2.0 and VAS will be administered as the primary outcome measures in addition to secondary outcome measures (speed and accuracy of minecraft).
  Interventions: Device: One Handed Video Game Controller Adapter

INTERVENTIONS:
Device: One Handed Video Game Controller Adapter — The one handed video game controller adapter was designed and 3D printed at Rehabilitation Centre for Children. It is a simple model that snaps onto an XBox One controller and uses a series of levers to allow access to almost all buttons of the controller from one side. There is both left and right sided versions

SUMMARY:
The goal of this clinical trial is to test a new one-handed video game controller adapter to determine if it helps improve how video games are played and enjoyed in children with an upper limb difference on one side. The main questions it aims to answer are:

* Is performance improved while playing video games with the adapter?
* Is user satisfaction or enjoyment improved while playing video games with the adapter?

Participants will:

* Answer questions about their limb difference and other demographics
* Be interviewed about their current and past video game playing experiences
* Learn how to use the adapter and have their performance with it evaluated
* Take the adapter home to use for 1 week, and be asked to record their experiences
* Have their performance with the adapter re-evaluated after a week of practice
* Be interviewed about their experience with the adapter

DETAILED DESCRIPTION:
Each participant will provide informed consent before participating in any study related activities. At initial evaluation, each participant will complete a demographic questionnaire, as well as a semi-structured interview about their previous video game playing experiences, and their motivation to participate in playing video games in the future. Following this interview, they will receive a training session from a team member on how to use the adapter and how to play Minecraft. This video game was chosen for its age appropriateness and need to use almost every button on the controller. Following the training, the investigators will collect initial outcome measure data for both the with and without adapter conditions.

Following the initial evaluation appointment, the participant will take home a tracking log, the video game controller adapter, and an Xbox with an Xbox One controller (if they do not already have one at home). Each participant will be asked to use the device daily and fill out the tracking log daily for 7 days. After which, each participant will return to RCC for the final evaluation appointment. At this time, outcome measurement will be repeated for gameplay with and without the adapter conditions. Finally, an exit semi-structured interview will be conducted to evaluate their experience with the adapter. Each participant will return the Xbox and controller if they were taken home. They will have the opportunity to keep the adapter if they wish.

ELIGIBILITY:
Inclusion Criteria:

* between the age of 7 and 17 years
* has a unilateral limb difference
* limb difference may be from any cause (congenital difference, traumatic loss, etc.)
* limb difference may be of any level (partial hand, wrist disarticulation, transradial, elbow disarticulation, transhumeral, shoulder disarticulation)
* ability to communicate in English
* cognitive ability to follow instructions
* eligible participants will be included regardless of history of prosthesis use
* lives locally (Winnipeg) or willing and able to travel to Rehabilitation Centre for Children for 2 appointments

Exclusion Criteria:

* less than 7 or greater than 17 years of age
* bilateral or no limb upper limb difference
* inability to communicate in English
* cognitive inability to follow instructions
* unable or unwilling to attend 2 appointments at Rehabilitation Centre for Children

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Quebec User Evaluation of Satisfaction with assistive Technology (QUEST 2.0) | Change in the QUEST (2.0) will be evaluated at baseline, and repeated one week later
  The QUEST 2.0 is an instrument designed to evaluate user satisfaction with a variety of assistive technologies. Each item in the measure is ranked by the participant on a scale of satisfaction (5 points from "not satisfied at all" to "very satisfied").
Visual Analog Scale (VAS) for Satisfaction (w/faces scale) | Change in satisfaction with play experience will be evaluated for both the with and without adapter conditions at baseline, and repeated one week later
  The VAS is a 10cm horizontal line, faces below it to indicate high to low satisfaction. The participant will mark how satisfied with their experience they are by placing an X on the corresponding position on the line.

SECONDARY OUTCOMES:
Time to complete obstacle course | Change in time to complete the obstacle course will be recorded for the with and without adapter condition at baseline and one week later
  A standardized video game based obstacle course will be performed in the with and without adapter condition. Time to complete in each condition will be recorded.
Errors to complete obstacle course | Change in errors to complete the obstacle course will be completed for the with and without adapter condition at baseline and one week later
  A standardized video game based obstacle course will be performed in the with and without adapter condition and errors in completion will be counted by an observer.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan C Guglich, C.P.(c), MSc., Principal Investigator — Rehabilitation Centre for Children
Locations (1):
- Rehabilitation Centre for Children, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jurdi S, Montaner J, Garcia-Sanjuan F, Jaen J, Nacher V. A systematic review of game technologies for pediatric patients. Comput Biol Med. 2018 Jun 1;97:89-112. doi: 10.1016/j.compbiomed.2018.04.019. Epub 2018 Apr 25. PMID 29715597
- [Background] Michielsen A, Van Wijk I, Ketelaar M. Participation and quality of life in children and adolescents with congenital limb deficiencies: A narrative review. Prosthet Orthot Int. 2010 Dec;34(4):351-61. doi: 10.3109/03093646.2010.495371. Epub 2010 Aug 13. PMID 20704518
- [Background] Granic I, Lobel A, Engels RC. The benefits of playing video games. Am Psychol. 2014 Jan;69(1):66-78. doi: 10.1037/a0034857. Epub 2013 Dec 2. PMID 24295515

DOCUMENTS (1):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT05981664/Prot_000.pdf